CLINICAL TRIAL: NCT07141654
Title: Empowering Families in Early Detection: Implementing Family-Led Recording for Early Diagnosis of Cerebral Palsy in Preterm Infants
Brief Title: This Study Aims to Evaluate the Validity of Family-led Recordings for General Movement Assessment (GMA) Compared to Provider-led Recording in Neonates Born Under 29weeks
Status: Not yet recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Jarred Garfinkle, Principal investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2026-11839
Record Dates: First submitted 2025-08-18; First posted 2025-08-26 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Cerebral Palsy; General Movement Assessment; Prematurity
MeSH Terms: conditions — Cerebral Palsy; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the validity of family-led recordings for General Movements Assessment (GMA) compared to provider-led recordings in neonates born <29 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Newborns < 29 weeks gestation admitted to the Montréal Children's hospital (MCH) Neonatal Intensive Care Unit (NICU), who are anticipated to be followed at the MCH Neonatal Follow-up Clinic
2. Parents can communicate in French or English
3. Intention to come for regular follow-up in the MCH Neonatal Clinic and/or Physical/Occupational therapy appointments

Exclusion Criteria:

* None

Max Age: 29 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborns < 29 weeks gestation admitted to the MCH NICU, who are anticipated to be followed at the MCH Neonatal Follow-up Clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Score at the Prechtl Qualitative General Movements Assessment | From enrollment up to the 18 months corrected age
  evaluate the validity of family-led recordings for General Movement Assessment (GMA) compared to provider-led recordings in neonates born <29 weeks using the Prechtl Qualitative General Movements Assessment

SECONDARY OUTCOMES:
Measure prognostic value using local Canadian Neonatal Network (CNN) and Canadian Neonatal Follow Up Network (CNFUN) databases and electronic medical chart review | From enrollment up to 18 months corrected age
  to measure the prognostic value of the GMA in predicting Cerebral Palsy(CP) at 18 months corrected age. Information on patient characteristics and outcomes will be collected from the local Canadian Neonatal Network (CNN) and Canadian Neonatal Follow Up Network (CNFUN) databases for all infants meeting inclusion criteria. Additional data around GMA and neurodevelopment not included in the CNN/CNFUN databases will be collected through electronic medical chart review of all infants meeting inclusion criteria.
Assess age at referral | From enrollment up to 18 months corrected age
  to assess the age at referral for community rehabilitation services for infants with GMA early signs of CP using patient electronic charts
Assess parental satisfaction using a feedback questionnaire | From enrollment up to 18 months corrected age
  to assess the parental satisfaction with the GMA administration process and the training materials provided using a feedback questionnaire